CLINICAL TRIAL: NCT00857662
Title: U.S. Multicenter, Randomized Controlled Study Comparing the Performance fo Onyx(EVOH) and TRUFILL® (n-BCA)in Presurgical Embolization of Brain Arteriovenous Malformations (BAVMs)
Brief Title: Study Comparing Onyx and TRUFILL in Brain Arteriovenous Malformations (AVMs)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medtronic Neurovascular Clinical Affairs (Industry)
Collaborators: Micro Therapeutics Inc. (Industry)
Responsible Party: Linda Simpson/Director of Clinical Affairs, Microtherapeutics, Inc dba ev3, Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G000296
Record Dates: First submitted 2009-03-05; First posted 2009-03-09 (Estimated); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Brain Arteriovenous Malformations
Keywords: US Multicenter; Randomized; Onyx; Brain Arteriovenous Malformation (BAVMs)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Onyx (Experimental)
  Interventions: Device: Onyx
- TRUFILL (Active Comparator)
  Interventions: Device: TRUFILL

INTERVENTIONS:
Device: Onyx — Embolization
  Arms: Onyx
Device: TRUFILL — Embolization
  Arms: TRUFILL

SUMMARY:
Test whether AVMs treated with Onyx is equivalent to treatment with n-BCA. Success is defined as an AVM size reduction greater than 50%

DETAILED DESCRIPTION:
Recent advances in the endovascular treatment of arteriovenous malformations (AVMs) have increased the number of patients with brain AVMs for whom embolization therapy may be appropriate. The permanency of obliterated nidi and occurrence of procedural complications are thought to be at least partially influenced by the characteristics of the material used, with liquid agents more likely to reach and occlude the AVM nidus compared to particulate embolic agents.

The only liquid embolic agent approved in the U.S. for the presurgical embolization of AVMs is TRUFILL®. TRUFILL n-butyl cyanoacrylate (n-BCA) is a liquid adhesive that polymerizes into a solid material upon contact with blood fluids or tissue, via an anionic mechanism. TRUFILL Ethiodized Oil is mixed into the n-BCA monomer as a radiopaque polymerizing retardant. TRUFILL Tantalum Powder may also be added for radiopacity. The TRUFILL n-BCA Liquid Embolic System received U.S. FDA premarket approval on September 25, 2000 (P990040) for use in the embolization of cerebral AVMs, when presurgical devascularization is desired.

Onyx™ is a non-adhesive liquid embolic agent comprised of ethylene vinyl alcohol (EVOH) copolymer dissolved in dimethyl sulfoxide (DMSO), and of micronized tantalum powder. Onyx precipitates into a solid on contact with blood fluids, due to rapid diffusion of the DMSO solvent. The Onyx Liquid Embolic System received the European "CE mark" in July 1999, and has been available outside of the U.S. since September 1999 for use in the embolization of AVMs.

The purpose of this randomized-controlled study is to obtain prospective clinical data on the performance of Onyx (investigational device) and TRUFILL (control device) in the presurgical embolization of brain AVMs. Device safety will be assessed by comparing overall and device-related morbidity and mortality. The primary efficacy endpoint is the angiographic reduction in AVM size (volume) achieved. The objective is to demonstrate that Onyx is no worse than TRUFILL within a specified clinical tolerance. Study results will be used to support a premarket approval application for Onyx in the presurgical embolization of brain AVMs.

ELIGIBILITY:
Inclusion Criteria:

* The patient or patient's guardian understands and will sign the informed consent for the procedure
* The patient has a confirmed diagnosis of a brain AVM in the cerebral cortex, cerebellum or dura mater as visualized by angiography or cross sectional imaging.
* The brain AVM has a Spetzler-Martin grade of I, II, III, or IV. If the brain AVM has a Spetzler-Martin grade of I or II, the anticipated benefit of embolization for surgical resection is greater than the risk of the embolization procedure (e.g., patient stability).
* The patient is a candidate for surgical resection of the AVM post embolization.
* The patient is clinically and neurologically stable, for a minimum of 24 hours prior to embolization.
* The patient agrees to have, and is capable of completing, all study-related exams and procedures.
* Patient of any age.

Exclusion Criteria:

* The patient is pregnant.
* The patient has a brain AVM with high flow arteriovenous fistulae that the investigator has determined to be unsuitable for embolization.
* The brain AVM has a Spetzler-Martin grade of V.
* The patient is participating in another research study involving another investigational device, procedure or drug.
* The brain AVM has been previously treated with another embolization agent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2001-05; Primary Completion 2003-04 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Angiographic reduction in AVM size (volume) of 50% or greater, where angiographic size reduction is defined as the change from the original AVM size prior to any embolization procedure, to the AVM size after the last embolization. | Post final embolization

SECONDARY OUTCOMES:
Safety will be assessed by the nature and severity of adverse events | 3 months post discharge
Surgical blood loss
Surgical resection time

CONTACTS AND LOCATIONS:
Overall Officials: Gary Duckwiler, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States